CLINICAL TRIAL: NCT03077386
Title: Enhancing Community Health Through Patient Navigation, Advocacy and Social Support
Acronym: ENCOMPASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Alberta Innovates Health Solutions (Other); Canadian Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: REB17-0360
Record Dates: First submitted 2017-03-01; First posted 2017-03-13 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Hypertension; Diabetes Mellitus, Type 2; Chronic Kidney Diseases; Ischemic Heart Disease; Congestive Heart Failure; Chronic Obstructive Pulmonary Disease; Asthma
Keywords: patient navigator; community health navigator; multi-morbidity; primary care; social determinants of health
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic; Myocardial Ischemia; Heart Failure; Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Intervention Model Description: The investigators will test the effectiveness of the ENCOMPASS program using a parallel, two-arm, pragmatic, wait-list control, cluster-randomized trial. Half the clinics will be randomized to receive the intervention immediately, serving as the intervention group, while the other half will receive the intervention after a 6 month waiting period, acting as control sites during their first 6 months. Once implemented, the ENCOMPASS program will remain available to clinics until the end of the funding period. Control patients will continue to receive usual care until their clinic becomes eligible for the program.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ENCOMPASS program (Experimental): Clinics assigned to the intervention will receive the ENCOMPASS intervention and a CHN will be matched to their clinic and be available to patients that meet the eligibility criteria.
  Interventions: Behavioral: ENCOMPASS Intervention
- Usual care (No Intervention): Patients not enrolled in the intervention will continue to receive care as usual until their clinic receives the intervention.

INTERVENTIONS:
Behavioral: ENCOMPASS Intervention — Patients will be matched to a CHN who will conduct a needs assessment to determine the frequency of meetings. A CHN may perform any of the following: providing information to a patient's health care provider, translation, advocating for the patient, connecting the patient with resources (i.e., social, financial, insurance), helping patients set health related goals, liaising with a patient's employer, facilitating health care referrals and appointments, monitoring appointments, and facilitating transportation to appointments. These activities may require the CHN to be physically present at appointments or have direct contact with the patient's health care provider. Goal setting and support will be provided in person or over the telephone using motivational interviewing principles
  Other Names: Community Health Navigation Services
  Arms: ENCOMPASS program

SUMMARY:
Some patients who have multiple long-term health conditions have significant challenges accessing needed services despite available primary care and social services resources. Patient navigation programs may help those with complex health conditions improve their care and outcomes and if delivered by community health navigators (CHNs) who have close community ties, these programs have the potential to reduce barriers to care and increase access to coordinated, person-centred care. The ENCOMPASS program aims to improve the care and health outcomes for high-risk patients by linking patients with chronic disease with a CHN to help them navigate the health system, facilitate communication between patients and providers, improve patients' understanding of their conditions and treatment plans, and support patients in their self-management. In Canada, patient navigation programs have not been well studied or broadly implemented in patients with chronic disease, making a comprehensive evaluation of ENCOMPASS important. This program has great potential to improve care for patients with chronic diseases in primary care.

DETAILED DESCRIPTION:
Although non-communicable chronic disease is the leading cause of death in Canada, many patients with chronic diseases do not receive guideline-recommended therapy for a variety of reasons. Lack of awareness of publicly funded programs, financial constraints, personal circumstances, language and cultural barriers make it challenging for patients to follow recommendations. ENCOMPASS is a patient navigation intervention, delivered by community health navigators (CHNs), that will improve patient-centred care and outcomes by: helping patients navigate the health system, facilitating communication between patients and providers, improving patient understanding of their conditions and treatment plans, connecting patients with community resources and supporting patient self-management.

The ENCOMPASS intervention is based on an extensive literature review, and was refined in consultation with patients, operational partners, front-line care providers, and local and provincial policy makers. A pilot study has informed implementation, recruitment and data collection methods. This study will implement and test the intervention using a pragmatic cluster-randomized trial with a concurrent qualitative study. The objectives of this study are to determine the effectiveness of patient navigation, delivered by CHNs, in patients with multiple chronic diseases on: a) emergency department visits and hospital admissions over 12 months (primary outcome), b) patient-reported outcome and experience measures, and c) disease-specific clinical outcomes, compared with usual care. Additional objectives focus on practical aspects including understanding the experience of care from the patient and CHN perspective and factors influencing the intervention's ability to improve care and outcomes.

The effectiveness of ENCOMPASS will be studied using a parallel, two-arm, pragmatic, wait-list control, cluster-randomized trial (cRCT) in 16 clusters, with a target size of 1600 patients with chronic disease. If additional funding is realized the trial will be expanded to include additional clusters. Primary care practices with ~5 full-time physicians will be the cluster units and small practices of 2-3 physicians may be combined into one cluster. Half of the clusters will be randomized to receive the program immediately (Early Phase clusters), while the other half will be required to wait 6 months (Late Phase clusters). Randomization will be concealed, computer-generated and stratified by practice size. Although patients and providers cannot be blinded to the intervention, end-point evaluation will be blinded. The primary outcome will be assessed using administrative health data, eliminating risk of assessor bias. Control patients will receive usual care until the intervention is implemented in their clinic, at which time they will be eligible for the ENCOMPASS program.

Patients will meet with a research assistant at baseline, 6 and 12 months, with an additional 18 month follow-up for control patients, to assess clinical data, including weight, blood pressure, and patient-reported measures. Other endpoints (i.e., through administrative and laboratory data) will be assessed at 6, 12, and 24 months. Once implemented, the ENCOMPASS program will remain available to clinic patients until the end of the program funding period, which may be extended subject to budget decisions and preliminary results. A concurrent qualitative study will provide contextual information and will be used to make program refinements in the Late Phase, the impacts of which will be explored in a comparative analysis.

ELIGIBILITY:
Inclusion Criteria:

≥ 18 years of age with two or more of the following:

* Poorly controlled hypertension (most recent systolic blood pressure > 160 mmHg);
* Poorly controlled diabetes (A1C > 9% on at least one occasion within the past year);
* Stage 3b or greater chronic kidney disease (estimated glomerular filtration rate < 45 mL/min/1.73m2 in past year);
* Established ischemic heart disease (at least one instance of a physician billing diagnosis with a relevant International Classification of Diseases, 9th Edition [ICD-9] code recorded in electronic medical record (EMR), or known to health care team);
* Congestive heart failure (at least one instance of a physician billing diagnosis with a relevant ICD-9 code recorded in EMR, or known to health care team);
* Chronic obstructive pulmonary disease OR Asthma with at least two visits in the past year (at least 2 instances of a physician billing diagnosis with a relevant ICD-9 code, or known to health care team).

Exclusion Criteria:

* patient unable to provide informed consent;
* patient residing in a long-term care facility;
* physician discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2024-03-03 (Actual)

PRIMARY OUTCOMES:
Acute care utilization | Up to 36 months
  All emergency department visits and hospital admissions

SECONDARY OUTCOMES:
Health-related quality of life | Up to 24 months
  EQ-5D-5L (Euroqol 5 dimension- 5 level instrument) administration
Disease-specific intermediate health outcomes (hypertension) | Up to 24 months
  Blood pressure based on primary data collection
Disease-specific intermediate health outcomes (diabetes) | Up to 24 months
  Hemoglobin A1c based on laboratory data
Disease-specific intermediate health outcomes (appropriate medication use) | Up to 24 months
  Use of a statin where indicated (according to chronic disease guidelines)
Disease-specific intermediate health outcomes (heart failure) | Up to 24 months
  Number exacerbations based on administrative data
Disease-specific intermediate health outcomes (chronic obstructive pulmonary disease and asthma) | Up to 24 months
  Number exacerbation based on administrative data
Patient activation | Up to 24 months
  Patient activation measure (PAM) administration via survey questionnaire
Patient experience with chronic illness care | Up to 24 months
  Patient assessment of chronic illness care (PACIC) administration via survey questionnaire
Primary care attachment | Up to 24 months
  Usual provider of care index (UPC) based on physician claims data
Physician experience | 6- and 12-months post-implementation
  Open-ended questions via semi-structured interview
Medication adherence | Up to 24 months
  Pharmaceutical information network (PIN) administrative data
Mortality | Up to 24 months
  All-cause mortality based on administrative data
Weight | Up to 24 months
  Weight based on primary data collection
Social support | Up to 24 months
  Social support based on Medical Outcomes Study Social Support Survey
Smoking status | Up to 24 months
  Current smoker Yes/No
Depression score | Up to 24 months
  Patient Health Questionnaire - 9 item administration via survey questionnaire (PHQ-9). 4 point scale to measure depression ranging from a positive outcome response (not at all) to negative outcome response (nearly everyday).
Anxiety score | Up to 24 months
  Generalized Anxiety Disorder - 7 item administration via survey questionnaire (GAD-7). 4 point scale to measure anxiety ranging from a positive outcome response (not at all) to negative outcome response (nearly everyday).
Program costs | Up to 24 months
  Total operational costs
Physician costs | Up to 24 months
  Physician claims costs
Acute care costs | Up to 24 months
  Costs for emergency department visits and hospital admissions, based on RIW methods

CONTACTS AND LOCATIONS:
Overall Officials: Kerry A McBrien, MD, MPH, Principal Investigator — University of Calgary
Locations (1):
- Mosaic Primary Care Network, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Public Health Agency of Canada. Chronic Disease and Injury Framework Quick Stats, 2016 Edition. Retreived from http://www.phac-aspc.gc.ca/publicat/hpcdp-pspmc/36-8/assets/pdf/ar-04-eng.pdf
- [Background] Saher, MN (2014). Report of the Auditor General of Alberta: Health- Chronic Disease Management. Edmonton, AB: Office of the Auditor General of Alberta.
- [Background] Fortin M, Bravo G, Hudon C, Vanasse A, Lapointe L. Prevalence of multimorbidity among adults seen in family practice. Ann Fam Med. 2005 May-Jun;3(3):223-8. doi: 10.1370/afm.272. PMID 15928225
- [Background] Bayliss EA, Bayliss MS, Ware JE Jr, Steiner JF. Predicting declines in physical function in persons with multiple chronic medical conditions: what we can learn from the medical problem list. Health Qual Life Outcomes. 2004 Sep 7;2:47. doi: 10.1186/1477-7525-2-47. PMID 15353000
- [Background] Condelius A, Edberg AK, Jakobsson U, Hallberg IR. Hospital admissions among people 65+ related to multimorbidity, municipal and outpatient care. Arch Gerontol Geriatr. 2008 Jan-Feb;46(1):41-55. doi: 10.1016/j.archger.2007.02.005. Epub 2007 Apr 2. PMID 17403548
- [Background] Fortin M, Lapointe L, Hudon C, Vanasse A, Ntetu AL, Maltais D. Multimorbidity and quality of life in primary care: a systematic review. Health Qual Life Outcomes. 2004 Sep 20;2:51. doi: 10.1186/1477-7525-2-51. PMID 15380021
- [Background] Manns BJ, Tonelli M, Zhang J, Campbell DJ, Sargious P, Ayyalasomayajula B, Clement F, Johnson JA, Laupacis A, Lewanczuk R, McBrien K, Hemmelgarn BR. Enrolment in primary care networks: impact on outcomes and processes of care for patients with diabetes. CMAJ. 2012 Feb 7;184(2):E144-52. doi: 10.1503/cmaj.110755. Epub 2011 Dec 5. PMID 22143232
- [Background] McAlister FA, Majumdar SR, Eurich DT, Johnson JA. The effect of specialist care within the first year on subsequent outcomes in 24,232 adults with new-onset diabetes mellitus: population-based cohort study. Qual Saf Health Care. 2007 Feb;16(1):6-11. doi: 10.1136/qshc.2006.018648. PMID 17301194
- [Background] Shah BR, Hux JE, Austin PC. Diabetes is not treated as a coronary artery disease risk equivalent. Diabetes Care. 2007 Feb;30(2):381-3. doi: 10.2337/dc06-1654. No abstract available. PMID 17259516
- [Background] Sirois C, Moisan J, Poirier P, Gregoire JP. Suboptimal use of cardioprotective drugs in newly treated elderly individuals with type 2 diabetes. Diabetes Care. 2007 Jul;30(7):1880-2. doi: 10.2337/dc06-2257. Epub 2007 Mar 23. No abstract available. PMID 17384345
- [Background] Supina AL, Guirguis LM, Majumdar SR, Lewanczuk RZ, Lee TK, Toth EL, Johnson JA. Treatment gaps for hypertension management in rural Canadian patients with type 2 diabetes mellitus. Clin Ther. 2004 Apr;26(4):598-606. doi: 10.1016/s0149-2918(04)90062-8. PMID 15189757
- [Background] Tonelli M, Bohm C, Pandeya S, Gill J, Levin A, Kiberd BA. Cardiac risk factors and the use of cardioprotective medications in patients with chronic renal insufficiency. Am J Kidney Dis. 2001 Mar;37(3):484-9. PMID 11228171
- [Background] Tonelli M, Gill J, Pandeya S, Bohm C, Levin A, Kiberd BA. Barriers to blood pressure control and angiotensin enzyme inhibitor use in Canadian patients with chronic renal insufficiency. Nephrol Dial Transplant. 2002 Aug;17(8):1426-33. doi: 10.1093/ndt/17.8.1426. PMID 12147790
- [Background] Toth EL, Majumdar SR, Guirguis LM, Lewanczuk RZ, Lee TK, Johnson JA. Compliance with clinical practice guidelines for type 2 diabetes in rural patients: treatment gaps and opportunities for improvement. Pharmacotherapy. 2003 May;23(5):659-65. doi: 10.1592/phco.23.5.659.32203. PMID 12741441
- [Background] Ronksley PE, Sanmartin C, Campbell DJ, Weaver RG, Allan GM, McBrien KA, Tonelli M, Manns BJ, Hennessy D, Hemmelgarn BR. Perceived barriers to primary care among western Canadians with chronic conditions. Health Rep. 2014 Apr;25(4):3-10. PMID 24744042
- [Background] Freeman HP. The history, principles, and future of patient navigation: commentary. Semin Oncol Nurs. 2013 May;29(2):72-5. doi: 10.1016/j.soncn.2013.02.002. No abstract available. PMID 23651676
- [Background] Walkinshaw E. Patient navigators becoming the norm in Canada. CMAJ. 2011 Oct 18;183(15):E1109-10. doi: 10.1503/cmaj.109-3974. Epub 2011 Sep 19. No abstract available. PMID 21930738
- [Background] Parker VA, Lemak CH. Navigating patient navigation: crossing health services research and clinical boundaries. Adv Health Care Manag. 2011;11:149-83. doi: 10.1108/s1474-8231(2011)0000011010. PMID 22908669
- [Background] Pedersen A, Hack TF. Pilots of oncology health care: a concept analysis of the patient navigator role. Oncol Nurs Forum. 2010 Jan;37(1):55-60. doi: 10.1188/10.ONF.55-60. PMID 20044339
- [Background] Wells KJ, Battaglia TA, Dudley DJ, Garcia R, Greene A, Calhoun E, Mandelblatt JS, Paskett ED, Raich PC; Patient Navigation Research Program. Patient navigation: state of the art or is it science? Cancer. 2008 Oct 15;113(8):1999-2010. doi: 10.1002/cncr.23815. PMID 18780320
- [Background] Fischer SM, Sauaia A, Kutner JS. Patient navigation: a culturally competent strategy to address disparities in palliative care. J Palliat Med. 2007 Oct;10(5):1023-8. doi: 10.1089/jpm.2007.0070. No abstract available. PMID 17985954
- [Background] Shlay JC, Barber B, Mickiewicz T, Maravi M, Drisko J, Estacio R, Gutierrez G, Urbina C. Reducing cardiovascular disease risk using patient navigators, Denver, Colorado, 2007-2009. Prev Chronic Dis. 2011 Nov;8(6):A143. Epub 2011 Oct 17. PMID 22005636
- [Background] Goff SL, Pekow PS, White KO, Lagu T, Mazor KM, Lindenauer PK. IDEAS for a healthy baby--reducing disparities in use of publicly reported quality data: study protocol for a randomized controlled trial. Trials. 2013 Aug 7;14:244. doi: 10.1186/1745-6215-14-244. PMID 23919671
- [Background] Scott LB, Gravely S, Sexton TR, Brzostek S, Brown DL. Examining the effect of a patient navigation intervention on outpatient cardiac rehabilitation awareness and enrollment. J Cardiopulm Rehabil Prev. 2013 Sep-Oct;33(5):281-91. doi: 10.1097/HCR.0b013e3182972dd6. PMID 23823904